CLINICAL TRIAL: NCT00937482
Title: A Phase 1 Study of AZD2171 and WBRT in Patients With Brain Metastases
Brief Title: Cediranib Maleate and Whole Brain Radiation Therapy in Patients With Brain Metastases From Non-Small Cell Lung Cancer
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Administratively complete.
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2013-00575; 09-089; U01CA062490 (NIH)
Record Dates: First submitted 2009-07-09; First posted 2009-07-13 (Estimated); Last update posted 2013-03-08 (Estimated); Status verified 2013-03

CONDITIONS: Male Breast Cancer; Stage IV Breast Cancer; Stage IV Melanoma; Stage IV Non-small Cell Lung Cancer; Stage IV Renal Cell Cancer; Stage IVA Colon Cancer; Stage IVA Rectal Cancer; Stage IVB Colon Cancer; Stage IVB Rectal Cancer; Tumors Metastatic to Brain
MeSH Terms: conditions — Breast Neoplasms, Male; Breast Neoplasms; Melanoma; Carcinoma, Non-Small-Cell Lung; Carcinoma, Renal Cell; Colonic Neoplasms; Rectal Neoplasms; Brain Neoplasms | interventions — cediranib

ARMS (1):
- Treatment (cediranib maleate and WBRT) (Experimental): Patients receive oral cediranib maleate on day 1. Patients undergo whole-brain radiotherapy 5 days a week for 3 weeks beginning on day 3. Treatment continues treatment in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: cediranib maleate; Radiation: whole-brain radiation therapy

INTERVENTIONS:
Drug: cediranib maleate — Given orally
  Other Names: AZD2171; Recentin
Radiation: whole-brain radiation therapy — Undergo whole-brain radiotherapy
  Other Names: WBRT; whole-brain radiotherapy

SUMMARY:
This phase I trial is studying the side effects and best dose of cediranib maleate when given together with whole brain radiation therapy in treating patients with brain metastases from non-small cell lung cancer. Cediranib maleate may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth or by blocking blood flow to the tumor. Radiation therapy uses high-energy x-rays and other types of radiation to kill cancer cells and shrink tumors. Giving cediranib maleate together with radiation therapy may kill more tumor cells

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the safety and tolerability (maximum tolerated dose, or MTD) of AZD2171 when combined with WBRT in patients with brain metastases.

SECONDARY OBJECTIVES:

I. To describe the objective response rate (ORR) in the central nervous system (CNS), neurologic progression-free survival (N-PFS), overall survival, and cause of death, and to explore the vascular normalization window using serial, noninvasive imaging parameters.

OUTLINE:

Patients receive oral cediranib maleate on day 1. Patients undergo whole-brain radiotherapy 5 days a week for 3 weeks beginning on day 3. Treatment continues treatment in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed periodically.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have one of the following histologically or cytologically confirmed cancers diagnosed no less than 12 weeks prior to study enrollment: non-small cell lung cancer, breast cancer, melanoma, colorectal cancer, or renal cell cancer
* Patients must have >= 1 radiologically proven (by gadolinium-enhanced [Gd-] MRI) parenchymal brain metastasis
* Patients must have had no prior therapy for brain metastases with the exception of craniotomy for resection of brain metastases within 8 weeks of study entry
* At least 2 weeks since last prior radiotherapy or chemotherapy (6 weeks if the last regimen included nitrosoureas, mitomycin C or bevacizumab)
* At least 4 weeks since last surgery
* There is no limit to the number of extracranial sites of disease
* Karnofsky performance status >= 70%
* Life expectancy of greater than 8 weeks
* Leukocytes >= 3,000/mcL
* Absolute neutrophil count >= 1,500/mcL
* Platelets >= 100,000/mcL
* Total bilirubin =< 1.5 x upper limit of reference range (ULRR)
* AST (SGOT)/ALT (SGPT) =< 2.5 x ULRR or =< 5 x ULRR for patients with liver metastases
* Creatinine =< 1.5 x ULRR or creatinine clearance >= 50 mL/min calculated by Cockcroft-Gault for patients with creatinine levels > 1.5 x ULRR
* Patients must have a mini-mental status exam (MMSE) score >= 15
* Women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation; women of child-bearing potential must have a negative pregnancy test prior to study entry; should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately
* Ability to understand and the willingness to sign a written informed consent document

Exclusion Criteria:

* Patients who have had chemotherapy or radiotherapy within 2 weeks (6 weeks for nitrosoureas, mitomycin C or bevacizumab) prior to entering the study or those who have not recovered from adverse events due to agents administered more than 2 weeks earlier
* Patients receiving any other investigational agents or who have participated in an investigational therapeutic trial within the past 30 days
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to AZD2171
* Patients taking enzyme-inducing antiepileptic drugs (EIAED); patients may be on non-enzyme-inducing antiepileptic drugs (NEIAED) or may be on no antiepileptic drugs (AED); patients off EIAED for >= 2 weeks are eligible
* Although the following medications are not contra-indicated on this study, each should be used with extreme caution, due to potential nephrotoxic effects: vancomycin, amphotericin, pentamidine
* Patients who have leptomeningeal disease as the only site of CNS involvement are excluded, because disease progression is difficult to evaluate and standard treatment options and the extent of radiation may differ
* Patients taking oral anticoagulant drugs are excluded; patients may be taking low molecular weight heparin
* Patients with a mean corrected QT interval > 470 milliseconds (with Bezett's correction) or patients with familial prolonged QT syndrome
* Patients with > 1+ proteinuria on two successive urine dipstick assessments taken no less than 7 days apart, unless urinary protein is < 1.5 g in a 24-hour period; if first urinalysis shows no protein, then a repeat urinalysis is NOT required
* Patients with significant hemorrhage (> 30mL bleeding per episode in previous 3 months) or hemoptysis (> 5mL fresh blood in previous 4 weeks)
* Patients who have brain imaging (CT or MRI) evidence of acute intra- or peri- tumoral hemorrhage > grade 1; patients with punctuate hemorrhage or hemosiderin deposition are eligible
* Patients who cannot undergo MRI safely
* Uncontrolled intercurrent illness including, but not limited to ongoing or active infection, uncontrolled hypertension (> 140 systolic or > 90 diastolic mm Hg), New York Heart Association class III or IV heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* Patients with conditions requiring concurrent drugs or biologics with proarrhythmic potential
* Pregnant women are excluded from this study; breastfeeding should be discontinued if the mother is treated with AZD2171
* HIV-positive patients on combination antiretroviral therapy are ineligible

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2009-08; Primary Completion 2011-03 (Actual)

PRIMARY OUTCOMES:
MTD defined as the dose at which no patients develop treatment-related grade 5 toxicity and less than 30% of patients develop acute dose limiting toxicities (DLT) assessed using NCI CTCAE version 4.0 | 7 weeks

SECONDARY OUTCOMES:
Objective response in the CNS | Up to 1.5 years
Neurologic progression-free survival | Time from start of treatment to time of progression in the CNS, assessed up to 1.5 years
  N-PFS will be summarized using a Kaplan-Meier survival curve.
Overall survival | From study entry until death due to any cause, assessed up to 1.5 years
  Overall survival will be summarized using a Kaplan-Meier survival curve.
Cause of death | Up to 1.5 years
  The proportion of patients who fall into each category will be tabulated.
Vascular MRI studies | Up to 1.5 years

CONTACTS AND LOCATIONS:
Overall Officials: April Eichler, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital Cancer Center, Boston, Massachusetts, United States